CLINICAL TRIAL: NCT06755164
Title: Effects of Combined Aerobic and Cognitive Training in a Simultaneous or Sequential Paradigm on Cognition and Brain Functional Activity in Patients with Amnesic Mild Cognitive Impairment
Brief Title: Effects of Combined Aerobic and Cognitive Training in a Simultaneous or Sequential Paradigm on Cognition and Brain Functional Activity in Patients with AMCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Prof., IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: aMCI SIM-SEQ
Record Dates: First submitted 2024-12-13; First posted 2025-01-01 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment (MCI); AMCI - Amnestic Mild Cognitive Impairment; Neurodegenerative Dementia; Neurodegenerative Disease
Keywords: Neurorehabilitation; cognitive training; aerobic training; combined training; cognitive rehabilitation; episodic memory; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Neurodegenerative Diseases | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: This study is a national, monocentric, double-blind, randomized, controlled, comparative, multi-parametric and parallel-group trial.
  Patients with a diagnosis of aMCI will be screened to establish eligibility for participation. Once enrolled, participants will be randomized through random.org software in the two experimental groups: 1) SIM (simultaneous) and 2) SEQ (sequential) aerobic-cognitive training. Allocation concealment will be carried out through closed and opaque mails by a blind operator. All patients will undergo the combined training for 3 months, with sessions scheduled twice a week, lasting 70 minutes each.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be maintained for allocation concealment, which will be carried out through closed and opaque mails by a blind operator. Patients will be labelled with a numerical code to ensure anonymisationPatients, assessors (neurologists, neuropsychologists and physiotherapists who will evaluate patient inclusion in the study) and statisticians will be blind to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SIM (simultaneous aerobic and cognitive training) (Experimental): In the SIMULTANEOUS Group (SIM), the aerobic and cognitive training will be performed simultaneously (i.e. the cognitive training will be performed during the aerobic training).
  Interventions: Other: Simultaneous aerobic and cognitive training (SIM)
- SEQ (sequential aerobic and cognitive training) (Experimental): In the SEQUENTIAL Group (SEQ), the aerobic and cognitive training will be performed sequentially (i.e. the cognitive training will follow the aerobic training).
  Interventions: Other: Sequential aerobic and cognitive training (SEQ)

INTERVENTIONS:
Other: Simultaneous aerobic and cognitive training (SIM) — The SIMULTANEOUS Group (SIM) will undergo15 minutes of stretching and preparatory mobilization + 40 minutes of cyclette (5 minutes warm-up, 30 minutes aerobic and cognitive training, 5 minutes cool-down) + 15 minutes of mobilization and deep breathing (total: 70 minutes). Patients will perform the cognitive training sited on the cyclette using an adapted computer screen and a joystick.
  Arms: SIM (simultaneous aerobic and cognitive training)
Other: Sequential aerobic and cognitive training (SEQ) — The SEQUENTIAL Group (SEQ) will undergo 40 minutes of cyclette (5 minutes warm-up, 30 minutes aerobic training, 5 minutes cool-down), + 30 minutes of cognitive training (total: 70 minutes). Patients will perform the cognitive training after the aerobic training, sited on a desk using a computer and a joystick.
  Arms: SEQ (sequential aerobic and cognitive training)

SUMMARY:
Mild Cognitive Impairment (MCI) is a condition in which patients show an objective evidence of impairment in one or more cognitive domains but a spared independence in daily functional abilities. The cognitive domain which results to be the most impaired defines the clinical subtype. Specifically, the amnestic subtype of MCI (aMCI), which is the most frequent, is characterised by deficits in episodic memory and visuospatial abilities. Current literature reports that prompt and focused rehabilitation provided early in the disease course might slow down the development of the neurodegenerative condition. The coupling between cognitive and aerobic trainings is the most incisive non-pharmacological treatment, and its effects have been demonstrated to have an impact on global cognitive functions, quality of life, aerobic capacity, and mood in the elderly with aMCI. However, the best modality for coupling aerobic and cognitive trainings (i.e., whether sequential-SEQ: aerobic training followed by cognitive training; or simultaneous-SIM: cognitive training during aerobic training) is still unknown. The aim of the present study is to determine which modality, among SEQ or SIM, is the most incisive training in patients with aMCI. Using a Randomized Controlled design, the effect of this combined aerobic-cognitive non-pharmachological training in both modalities will be evaluated on cognitive changes assessed with standard and computerized neuropsychological batteries and in functional activity during a task-based functional Magnetic Resonance Imaging (fMRI) scan.

DETAILED DESCRIPTION:
This study will be the first one aimed at investigating the effects of a combined aerobic and cognitive training in the two different paradigms (SIM and SEQ) on cognitive functioning and brain functional MRI activity in patients with aMCI. Previous studies on aMCI patients reported that the combination of cognitive and aerobic training is more effective than the single treatments alone on both clinical and MRI outcome measures. Specifically, with the proposed training we expect to obtain ameliorative effects in terms of episodic memory, visuospatial abilities, cerebral activity and aerobic capacities, with a consequent benefit on quality of life and mood in both experimental groups; in addition, we also expect a reduction of IL-6 and TNF-alpha expression levels, and an enhancement of the BDNF.

The combined aerobic-cognitive training (in SIM and SEQ modalities) will have a duration of 3 months, with 24 sessions scheduled twice a week for 70 minutes each.

The first session will last 10 minutes more compared to the others in order to provide participants with all information concerning the cognitive task that they will perform during (in SIM condition) or after the aerobic training (in SEQ condition).

Aerobic and cognitive exercises will be the same for both groups (SIM and SEQ) and will be characterized as follows:

* Aerobic training: 30 minutes of cyclette at 40-59% heart rate reserve (HRR) or 64-76% maximum heart rate (corresponding at Rating of Perceived Exertion by Borg -BORG RPE= 12-13 -moderate intensity-).16 The cardiac frequency will be monitored by pulse oxymeter.
* Cognitive training: the entire training will last for 30 minutes and will consist of two cycles of a memory task (lasting 10 minutes) and a visuospatial task (5 minutes).

For the SIM condition, patient will perform the cognitive training sited on the cyclette using an adapted computer screen and a joystick.

For the SEQ condition, patient will perform the cognitive training sited on a desk using a computer and a joystick.

The aerobic training will be performed on a cyclette. For the cognitive training, the cognitive exercises will train two cognitive domain 1) memory and 2) visuospatial function. 1) During the mnemonic exercises, the patients will be asked to observe a screen on which different stimuli (objects) will be presented and to remember all of them. Then the subjects will be asked to recall the most of the observed objects. The number of stimuli (objects) will progressively increase in order to progressively improving the difficulty of the mnemonic training. 2) The visuospatial task will consist on the navigation in a labyrinth projected onto a screen. The subjects will have a mouse/joystick with which they will move through the labyrinth in order to find the shortest way to exit.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of amnesic mild cognitive impairment according to the current diagnostic criteria;
* age>60 years;
* stable acetylcholinesterase inhibitors and/or memantine at the time of enrolment for at least one month;
* subscription of the consent for personal data treatment and patients' informed consent for participation in the present study.

Exclusion Criteria:

* patients with a history of other systemic, neurologic, psychiatric diseases, head injury, cardiovascular events, and cerebrovascular alterations visible at an MRI scan;
* patients with a family history of neurodegenerative disorders;
* patients with a history of alcohol and/or psychotropic drugs abuse;
* patients who are used to do regular physical and/or cognitive activity;
* contraindication to perform MRI scan (cardiac pace-maker or other types of cardiac catheters, splinters or metallic shards, metallic prosthesis not compatible with magnetic field generated by MRI, claustrophobia, pregnancy, breastfeeding).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Episodic memory improvement | Baseline, month 3, month 9
  The primary aim of the study is to investigate episodic memory improvement (investigated with changes in the Alzheimer's Disease Assessment Scale (ADAS-cog scale), both in short- (sooner after training) and in long-term (6 months after training). ADAS-Cog scale is a useful tool which is widely employed to assess global cognitive functioning in patients with several neurodegenerative conditions including MCI. Range score is from 0 to 70. Lower scores indicate better performance.

SECONDARY OUTCOMES:
Functional MRI changes | Baseline, month 3
  Modifications in cerebral functional activity, measured through BOLD signal, soon after training using a task-based fMRI approach.
Changes in submaximal aerobic/functional walking capacity | Baseline, month 3, month 9
  The 6-minute walking test (6MWT) measures the distance a subject walks in 6 minutes and is used to assess changes in performance capacity
Mood changes | Baseline, month 3, month 9
  Changes in mood, as measured by the Beck Depression Inventory (BDI), following treatment at both short- and long-term follow-up. BDI is a 21-item, self-administered questionnaire designed to assess the severity of respondents' depression during the weeks prior to completing the questionnaire.
Quality of life changes | Baseline, month 3, month 9
  Modifications in quality of life as measured by the 12-item Short Form Survey (SF-12) after treatment at the short- and long-term follow up. The SF-12 is a 12-questions instrument for assessing self-reported health-related quality of life.
Inflammatory cytokines changes | Baseline, month 3, month 9
  To observe a reduction in inflammatory cytokines expression levels, specifically in interleukin-6 (IL-6) and tumor necrosis factor-α (TNF-alpha) levels, measured at the short- and long-term follow up. This biochemical effects will have a positive effect on brain-derived neurotrophic factor (BDNF).
Correlation between BOLD activity during task-based fMRI and after-treatment changes in cognition | month 3, month 9
  Correlation between fMRI BOLD activity and changes in cognitive function in both conditions (SIM and SEQ) after treatment at short and at long-term follow up.
Correlation between after-treatment changes in BOLD fMRI activity and cognition | Month 3
  Correlation between changes in BOLD activity and cognitive functioning in both conditions (SIM and SEQ) after treatment at short and at long-term follow up.
Correlation between biological factors and after-treatment changes in cognition | Baseline, month 3, month 9
  Correlation between changes in cognitive functioning and biological factors in both conditions (SIM and SEQ) after treatment at short and at long-term follow up.
Differences in patterns of brain activation between HC and patients | Baseline
  To study brain activation differences between patients and healthy subjects by comparing fMRI BOLD activity.
Cognitive differences between HC and patients | Baseline
  Baseline cognitive differences between patients and healthy subjects using the Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-Cog scale).
Biological differences between HC and patients | Baseline
  Biological differences in BDNF, IL-6, and TNF-alpha levels between patients and healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Lam LC, Chan WC, Leung T, Fung AW, Leung EM. Would older adults with mild cognitive impairment adhere to and benefit from a structured lifestyle activity intervention to enhance cognition?: a cluster randomized controlled trial. PLoS One. 2015 Mar 31;10(3):e0118173. doi: 10.1371/journal.pone.0118173. eCollection 2015. PMID 25826620
- [Background] Perneczky R, Pohl C, Sorg C, Hartmann J, Tosic N, Grimmer T, Heitele S, Kurz A. Impairment of activities of daily living requiring memory or complex reasoning as part of the MCI syndrome. Int J Geriatr Psychiatry. 2006 Feb;21(2):158-62. doi: 10.1002/gps.1444. PMID 16416470
- [Background] Train the Brain Consortium. Randomized trial on the effects of a combined physical/cognitive training in aged MCI subjects: the Train the Brain study. Sci Rep. 2017 Jan 3;7:39471. doi: 10.1038/srep39471. PMID 28045051
- [Background] Suo C, Singh MF, Gates N, Wen W, Sachdev P, Brodaty H, Saigal N, Wilson GC, Meiklejohn J, Singh N, Baune BT, Baker M, Foroughi N, Wang Y, Mavros Y, Lampit A, Leung I, Valenzuela MJ. Therapeutically relevant structural and functional mechanisms triggered by physical and cognitive exercise. Mol Psychiatry. 2016 Nov;21(11):1633-1642. doi: 10.1038/mp.2016.19. Epub 2016 Mar 22. PMID 27001615
- [Background] Baglio F, Griffanti L, Saibene FL, Ricci C, Alberoni M, Critelli R, Villanelli F, Fioravanti R, Mantovani F, D'amico A, Cabinio M, Preti MG, Nemni R, Farina E. Multistimulation group therapy in Alzheimer's disease promotes changes in brain functioning. Neurorehabil Neural Repair. 2015 Jan;29(1):13-24. doi: 10.1177/1545968314532833. Epub 2014 Apr 29. PMID 24788581
- [Background] Stigger FS, Zago Marcolino MA, Portela KM, Plentz RDM. Effects of Exercise on Inflammatory, Oxidative, and Neurotrophic Biomarkers on Cognitively Impaired Individuals Diagnosed With Dementia or Mild Cognitive Impairment: A Systematic Review and Meta-Analysis. J Gerontol A Biol Sci Med Sci. 2019 Apr 23;74(5):616-624. doi: 10.1093/gerona/gly173. PMID 30084942
- [Background] Canu E, Sarasso E, Filippi M, Agosta F. Effects of pharmacological and nonpharmacological treatments on brain functional magnetic resonance imaging in Alzheimer's disease and mild cognitive impairment: a critical review. Alzheimers Res Ther. 2018 Feb 20;10(1):21. doi: 10.1186/s13195-018-0347-1. PMID 29458420
- [Background] Anderson-Hanley C, Barcelos NM, Zimmerman EA, Gillen RW, Dunnam M, Cohen BD, Yerokhin V, Miller KE, Hayes DJ, Arciero PJ, Maloney M, Kramer AF. The Aerobic and Cognitive Exercise Study (ACES) for Community-Dwelling Older Adults With or At-Risk for Mild Cognitive Impairment (MCI): Neuropsychological, Neurobiological and Neuroimaging Outcomes of a Randomized Clinical Trial. Front Aging Neurosci. 2018 May 4;10:76. doi: 10.3389/fnagi.2018.00076. eCollection 2018. PMID 29780318
- [Background] McEwen SC, Siddarth P, Rahi B, Kim Y, Mui W, Wu P, Emerson ND, Lee J, Greenberg S, Shelton T, Kaiser S, Small GW, Merrill DA. Simultaneous Aerobic Exercise and Memory Training Program in Older Adults with Subjective Memory Impairments. J Alzheimers Dis. 2018;62(2):795-806. doi: 10.3233/JAD-170846. PMID 29480182
- [Background] Karssemeijer EGA, Aaronson JA, Bossers WJ, Smits T, Olde Rikkert MGM, Kessels RPC. Positive effects of combined cognitive and physical exercise training on cognitive function in older adults with mild cognitive impairment or dementia: A meta-analysis. Ageing Res Rev. 2017 Nov;40:75-83. doi: 10.1016/j.arr.2017.09.003. Epub 2017 Sep 12. PMID 28912076
- [Background] Kavirajan H, Schneider LS. Efficacy and adverse effects of cholinesterase inhibitors and memantine in vascular dementia: a meta-analysis of randomised controlled trials. Lancet Neurol. 2007 Sep;6(9):782-92. doi: 10.1016/S1474-4422(07)70195-3. PMID 17689146
- [Background] Versijpt J. Effectiveness and cost-effectiveness of the pharmacological treatment of Alzheimer's disease and vascular dementia. J Alzheimers Dis. 2014;42 Suppl 3:S19-25. doi: 10.3233/JAD-132639. PMID 25061049
- [Background] Wimo A, Guerchet M, Ali GC, Wu YT, Prina AM, Winblad B, Jonsson L, Liu Z, Prince M. The worldwide costs of dementia 2015 and comparisons with 2010. Alzheimers Dement. 2017 Jan;13(1):1-7. doi: 10.1016/j.jalz.2016.07.150. Epub 2016 Aug 29. PMID 27583652
- [Background] Gauthier S, Reisberg B, Zaudig M, Petersen RC, Ritchie K, Broich K, Belleville S, Brodaty H, Bennett D, Chertkow H, Cummings JL, de Leon M, Feldman H, Ganguli M, Hampel H, Scheltens P, Tierney MC, Whitehouse P, Winblad B; International Psychogeriatric Association Expert Conference on mild cognitive impairment. Mild cognitive impairment. Lancet. 2006 Apr 15;367(9518):1262-70. doi: 10.1016/S0140-6736(06)68542-5. PMID 16631882
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249